CLINICAL TRIAL: NCT06926530
Title: Navigating Herbs and Supplements in Breast Cancer: Usage, Impact, and Personalized Approaches for Diverse Populations
Brief Title: Herbs & Supplements in Breast Cancer Usage, Impact, and Personalized Approaches for Diverse Populations
Status: Not yet recruiting | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE8124
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Breast Carcinoma
Keywords: Complementary and Alternative Medicine; Alternative medicine; Herbs; Supplements; Complementary therapies; Holistic health
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Participants will complete a one-time 33-question survey. The survey is comprised of three sections: (1) Section A includes 12 questions related to demographic information, (2) Section B consists of 2 questions addressing treatment characteristics, & (3) Section C contains 19 questions focusing on supplement usage.

SUMMARY:
This research study is enrolling participants diagnosed with breast cancer and receiving/received chemotherapy and/or endocrine therapy. The study's primary objective is to assess the differences in the use of herbs and supplements among the populations served at Cleveland Clinic Florida and Ohio by administering a participant-reported questionnaire.

DETAILED DESCRIPTION:
The world has seen a rise in the use of Complementary and Alternative Medicine (CAM) since the early 1980s. This interest in CAM was significant in the United States to the extent that Congress established and set the Dietary Supplement Health and Education Act of 1994 to define what a dietary supplement entails and to launch a legal framework that oversees these products. In 2020, the National Health and Nutrition Examination survey found that the prevalence of dietary supplements among adults was around 58.5%, with sales reaching $55.7 Billion. Notably, the consumption of dietary supplements is not limited to healthy individuals. Individuals with cancer are significant consumers of such products, with a prevalence rate as high as 50% in the United States. CAM use originates from traditional and cultural practices outside of the Western healthcare system. The literature on the association between CAM use and ethnicity presents conflicting data. Most of the available studies are old, dating to the early 2000s, and lack proper ethnic representation. Additionally, there is a notable gap in the literature regarding the utilization of CAM in breast cancer patients within ethnic minorities. This study aims to evaluate ethnicity and its influence on the use of herbs and supplements in early-stage breast cancer (Stages 1,2,3) in two populations: participants receiving care at Cleveland Clinic Florida and those receiving care at Cleveland Clinic Ohio. The investigators also aim to evaluate the interactions between the most used herbs and supplements with standard therapy, be it endocrine therapy or chemotherapy. The investigators will select the top 10 by frequency of the used herbs and supplements and cross-match it with the Memorial Sloan Kettering Cancer Center integrative medicine "Search about Herbs" (https://www.mskcc.org/cancer-care/diagnosis-treatment/symptom-management/integrative-medicine/herbs/search) as well as "Herbs at glance" via the NIH website (https://www.nccih.nih.gov/health/herbsataglance). Moreover, the investigators aim to determine the prevalence of herbs and supplements use in individuals with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older.
* Breast cancer diagnosis at pathologic stage (I, II, and III)
* Participants with regional lymph node involvement
* Received Chemotherapy and/ or Endocrine therapy
* Established patients followed by a medical oncologist at Cleveland Clinic Florida and Ohio
* Able and willing to participate in the one-time survey.

Exclusion Criteria:

* Under 18 years of age
* Prior history of cancer diagnosis
* Unable or unwilling to participate in the survey
* Distant Metastatic Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Established stages I, II, and III breast cancer patients at Cleveland Clinic Florida and Ohio who received care will be screened by the research fellow before or after their oncology visit.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Influence of ethnicity on herb/supplement usage among early stage breast cancer participants. | 5 months
  Univariate analysis in which Chi-square test or Fisher's exact test will be performed.

SECONDARY OUTCOMES:
Determine the ten most common herbs and supplements by frequency of use in each Cancer Center. | 5 months
Determine the Prevalence of Herbs and Supplements in breast cancer patients. | 5 months
Assess potential associations between Conventional treatments and Herbs/Supplements. | 5 months
  Measured by multiple logistic regression model
Association between cancer stage and herbs/supplement usage. | 5 months
  Measured by multiple logistic regression model

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stone, MD, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic Florida
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic Main Campus, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No